CLINICAL TRIAL: NCT02044237
Title: Decoupling as Internet Based Intervention: an Randomized Controlled Study to Treat Trichotillomania
Brief Title: Online Treatment of Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Novartis (Industry); Julia Bangerter-Rhyner Foundation Bale switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TTM
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Trichotillomania; Alexithymia; Quality of Life
Keywords: trichotillomania; online therapy
MeSH Terms: conditions — Trichotillomania; Affective Symptoms | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decoupling (Experimental): specific technic to reduce hair pulling
  Interventions: Behavioral: Decoupling
- progressive muscle relaxation (Active Comparator): Progressive relaxation relaxation technic
  Interventions: Behavioral: Progressive relaxation

INTERVENTIONS:
Behavioral: Decoupling
  Arms: Decoupling
Behavioral: Progressive relaxation
  Arms: progressive muscle relaxation

SUMMARY:
Online study for patients with trichotillomania. 4 main hypothesis.

1. Alexithymia and Trichotillomania correlated and regression analyses find association between them
2. we will be able to find patient who have never been treated before. Those will suffer to the same amount as previously treated patients
3. Decoupling will be more helpful than progressive muscle relaxation
4. different constructs of emotion regulation will show different trait and state characteristics in patients with trichotillomania

DETAILED DESCRIPTION:
Randomized controlled trial with about 100 participants.

ELIGIBILITY:
Inclusion Criteria:

* suffering from trichotillomania 18 to 65 years old

Exclusion Criteria:

* current drug or alcohol addiction current psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Severity of trichotillomania | 7 months

SECONDARY OUTCOMES:
alexithymia | 7 months

OTHER OUTCOMES:
Quality of life | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rufer, MD, Prof, Principal Investigator — University of Zurich
Locations (1):
- University of, Zurich, Switzerland

REFERENCES:
- [Background] Moritz S, Treszl A, Rufer M. A randomized controlled trial of a novel self-help technique for impulse control disorders: a study on nail-biting. Behav Modif. 2011 Sep;35(5):468-85. doi: 10.1177/0145445511409395. Epub 2011 Jun 8. PMID 21659318
- See also: affective regualation in trichotillomania - publication — http://www.ncbi.nlm.nih.gov/pubmed/26783728
- See also: randomized therapy study for trichotillomania- publication — http://www.ncbi.nlm.nih.gov/pubmed/26398632
- See also: alexithymia in trichotillomania - publication — http://www.ncbi.nlm.nih.gov/pubmed/24768249